CLINICAL TRIAL: NCT00672724
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Subjective Response to Treatment With Ramelteon in Adult Subjects With Chronic Insomnia by Utilizing an Interactive Voice Response System (IVRS) for Collecting Diary Data
Brief Title: Efficacy of Ramelteon in Adults With Chronic Insomnia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Issues with data collection tool
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-04-TL-375-041; U1111-1114-2738 (Registry Identifier: WHO)
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Chronic Insomnia
Keywords: Insomnia; Sleep Disorder; Drug Therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ramelteon 8 mg QD (Experimental)
  Interventions: Drug: Ramelteon
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon — Ramelteon 8 mg tablets, taken orally, once daily for up to 2 weeks.
  Other Names: Rozerem™; TAK-375
  Arms: Ramelteon 8 mg QD
Drug: Placebo — Ramelteon placebo-matching tablets, taken orally, once daily for up to 2 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate subjectively reported treatment effects of ramelteon, once daily (QD), in adults with chronic insomnia.

DETAILED DESCRIPTION:
Insomnia is characterized by difficulties initiating and maintaining sleep, or complaints of non-restorative and non-refreshing sleep. Transient insomnia affects approximately one-third to one-half of the US population, based on the results of 2 surveys of representative samples of the adult US population conducted by the Gallup Organization in which respondents were asked if they had "ever had difficulty sleeping." Based on reports of "regular" or "frequent" sleep difficulty, results from the same studies suggest that approximately one-tenth of the US population experiences chronic insomnia. The ideal treatment for insomnia would reduce the latency to onset of sleep and increase total sleep time, without a negative impact on sleep architecture and without safety concerns or next-day effects.

Ramelteon is under global development by Takeda Chemical Industries, Ltd., for the treatment of transient and chronic insomnia and for the treatment of Circadian Rhythm Sleep Disorders.

This study is being conducted to assess the treatment effects of ramelteon in adults through the use of daily entry of information into an interactive voice response system. Study participation in this study is anticipated to be about 1 month.

ELIGIBILITY:
Inclusion Criteria

* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Has had primary chronic insomnia as defined by Diagnostic and Statistical Manual of Mental Disorders, 4th Edition Revised for at least 3 months.
* Reports a history of subjective sleep latency greater than or equal to 60 min and a subjective total sleep time less than 6.5 hours.
* Habitual bedtime is between 10:00 PM and 1:00 AM.
* Willing to have a fixed bedtime and agrees to go to bed within plus or minus 30 minutes of the habitual bedtime during the entire study.
* Consistent access to a touch tone phone and are willing to complete telephone questionnaires twice daily during participation in the study.
* Willing to remain in bed for at least 6.5 hours each night during the entire study.
* Used pharmacological assistance to sleep 0-4 times per week in the last 3 months.
* Must complete the morning questionnaire on at least 4 of the first 7 mornings after Screening Visit 1.
* On at least 3 of the first 5 nights of single-blind placebo treatment, the subject must have a subjective sleep latency of greater than or equal to 45 minutes.
* On at least 3 of the first 5 nights of single-blind placebo treatment, the subject must have a subjective total sleep time of less than 6.5 hours.

Exclusion Criteria

* Known hypersensitivity to ramelteon or related compounds, including melatonin, and 5-hydroxytryptophan.
* Participated in any other investigational study and/or took any investigational drug within 30 days prior to the first dose of single-blind study medication.
* Sleep schedule changes required by employment (eg, shift worker) within 3 months prior to the first night of single-blind study medication.
* Has flown across greater than 3 time zones within 7 days prior to screening, or will travel across 2 or more time zones during the course of the study.
* Participated in a weight loss program or has substantially altered exercise routine within 30 days prior to the first night of singleblind study medication.
* Ever had a history of seizures, sleep apnea, and/or chronic obstructive pulmonary disease.
* History of psychiatric disorder within the past 6 months.
* History of fibromyalgia.
* History of drug addiction or drug abuse within the past 12 months.
* History of alcohol abuse within the past 12 months, as defined in Diagnostic and Statistical Manual of Mental Disorders, 4th Edition Revised and/or regularly consumes more than 2 alcoholic drinks per day.
* Current significant hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, hematologic, or metabolic disease, unless currently controlled and stable with protocol-allowed medication, within 30 days prior to the first night of single-blind study medication.
* Uses tobacco products or any other products that may interfere with the sleep wake cycle during nightly awakenings.
* Any clinically important abnormal finding as determined by a medical history, physical examination, electrocardiogram, or clinical laboratory tests, as determined by the investigator.
* Positive hepatitis panel.
* Any additional condition(s) that in the Investigator's opinion would:

  * affect sleep/wake function
  * prohibit the subject from completing the study
  * indicate that continuation in the study would not be in the best interests of the subject.
* Is required to take or continues taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication, including:

  * Anxiolytics
  * Central nervous system active drugs
  * Hypnotics
  * Narcotic analgesics
  * Antidepressants
  * Beta blockers
  * Anticonvulsants
  * St. John's Wort
  * Sedating H1 antihistamines
  * Kava-kava
  * Systemic steroids
  * Ginkgo-biloba
  * Respiratory stimulants
  * Over-the-counter and prescriptions stimulants
  * Decongestants
  * Over-the-counter and prescription diet aids
  * Antipsychotics
  * Melatonin and all other drugs or supplements known to affect sleep/wake

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1081 (Actual)
Dates: Start 2005-02; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Mean Subjective Sleep Latency determined through subject responses on morning questionnaire. | Day 8

SECONDARY OUTCOMES:
Mean Subjective Sleep Latency. | Day 15
Mean Subjective Total Sleep | Day 8
Mean Subjective Total Sleep | Day 15
Adverse Events. | Days 1, 8, and 15 or Final Visit.
Clinical Laboratory Tests Hematology | Day 15 or Final Visit.
Clinical Laboratory Tests Chemistry. | Day 15 or Final Visit.
Clinical Laboratory Tests Urinalysis | Day 15 or Final Visit.
Vital Signs. | Days 8 and 15 or Final Visit.
Electrocardiograms. | Day 15 or Final Visit.
Physical Examinations. | Day 15 or Final Visit.

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science, Study Director — Takeda
Locations (43):
- United States (43):
  - Mesa, Arizona
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Hot Springs, Arkansas
  - Cerritos, California
  - La Jolla, California
  - La Mesa, California
  - Oakland, California
  - Denver, Colorado
  - Bay Harbor Island, Florida
  - Brandon, Florida
  - Clearwater, Florida
  - DeLand, Florida
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Hollywood, Florida
  - Miami, Florida
  - Pembroke Pines, Florida
  - Pinellas Park, Florida
  - Vero Beach, Florida
  - Atlanta, Georgia
  - Austell, Georgia
  - Macon, Georgia
  - Boise, Idaho
  - Northbrook, Illinois
  - Prairie Village, Kansas
  - Wichita, Kansas
  - Louisville, Kentucky
  - Frederick, Maryland
  - Moorestown, New Jersey
  - Menlius, New York
  - New York, New York
  - Williamsville, New York
  - Salem, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Mogadore, Ohio
  - Philadelphia, Pennsylvania
  - Bristol, Tennessee
  - Chattanooga, Tennessee
  - Dallas, Texas
  - Fairfax, Virginia
  - Tacoma, Washington

REFERENCES:
- See also: Rozerem Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ROZEREMPI